CLINICAL TRIAL: NCT03889834
Title: Modification of Biological Parameters After Autologous Blood Transfusion of a Small Volume of Packed Red Blood Cells (200 Ml) in Healthy Volunteers
Brief Title: Biological Parameters Changes After Autologous Blood Transfusion of Red Blood Cells (200 Ml) in Healthy Volunteers.
Acronym: AUTOT-SPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoire antidopage français (LADF) (Unknown); World Anti-Doping Agency (Other); GR-Ex executive comitee (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: K180405J
Record Dates: First submitted 2019-02-18; First posted 2019-03-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: The Focus is on the Detection of the Consequences of Autologous Blood Transfusion in Healthy Volunteers
Keywords: autologous transfusion; doping; blood markers; detection
MeSH Terms: interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Autotransfusion: blood stored at 4 ° C (Experimental): Intervention: Autologous Blood Transfusion of packed red blood cells (200 ml) stored at 4 ° C for 31 days
  Interventions: Procedure: Autologous Blood Transfusion
- Autotransfusion: blood stored at -80°C (Experimental): Intervention: Autologous Blood Transfusion of packed red blood cells (200 ml) stored at -80°C for 31 days
  Interventions: Procedure: Autologous Blood Transfusion
- Controls not transfused (Other): no transfusion
  Interventions: Other: No transfusion

INTERVENTIONS:
Procedure: Autologous Blood Transfusion — Autotransfusion of packed red blood cells (200 ml) stored at 4 or -80°C for 31 days
  Arms: Autotransfusion: blood stored at -80°C; Autotransfusion: blood stored at 4 ° C
Other: No transfusion — no transfusion
  Arms: Controls not transfused

SUMMARY:
The purpose of this study is to evaluate if differences between samples of subjects obtained before autologous blood transfusion or samples of non-transfused subjects and samples of subjects after autologous blood transfusion can be identified. Analyses performed will focus on the morphological and biochemical parameters of red blood cells and associated microparticles. The final goal would be to find markers of autologous blood transfusion, that could be used to identify such doping practice.

DETAILED DESCRIPTION:
Methodology and study design:

Pr Olivier Hermine, coordinator of the laboratory of Excellence GR-EX regrouping EFS (Etablissement Français du Sang) and INSERM (Institut National de la Santé et de la Recherche Médicale) partners, and leader of the Centre d'Investigation Clinique (CIC) Necker (Hospital Necker, Paris, France) will assure the promotion of the clinical study for Paris Hospital consortium AP-HP (assistance Publique-Hôpitaux de Paris).

To reproduce two potential scenarios of autologous transfusion by an athlete, 1 bag of blood packed red blood cells (after leuko deprivation and centrifugation) will be either stored at 4°C or frozen at -80°C after addition of 40% w/v glycerol. Reinfusion will be performed 31 days later.

A clinical randomized double-blinded two-phase study will be conducted. Volunteers will be separated in 3 groups:

* Group 1: Volunteers with regular sports activities without Autologous Blood Transfusion (ABT)T (n=10)
* Group 2: Volunteers with regular sports activities receiving a 200ml ABT with refrigerated blood (n=10)
* Group 3: Volunteers with regular sports activities receiving a 200ml ABT with frozen blood (n=10)

To ensure volunteers safety, collection, preparation and pretransfusion blood testing will be performed by EFS (Versailles, France). ABT as well as collection of samples will be performed at the CIC Necker (Paris, France). Blood samples will be collected before blood removal, the day of the ABT just before reinfusion and after 3 hours, 8 hours, 24 hours and 48 hours post-ABT. To perform all the experiments 25ml blood (4x 5 ml BD Vacutainer EDTA tubes) will be taken at each time point:

1 will be dispatched to the French anti-doping laboratory (LADF) for haematological analysis (Orsay, France), 2 to the EFS (Créteil, France) for RBC and MPs morphological characterization and quantification (using antigen markers, band 3 on the surface of MPs), 2 to INTS for MPs isolation, characterization (band 3 on the surface of MPs and RBC) and for proteomic analysis and Western-Blot.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 35 years old
* Without health problem nor disease requiring regular medical treatment
* Free from any intercurrent acute pathology over 7 days
* Healthy volunteers who have regularly sport activity, able to have blood sample and is out-of-competition during the research
* Subject who did not practice a competition (or exhaustive training ) 3 days before the blood sample and the autotransfusion
* Affiliated to a social security regimen

Exclusion Criteria:

* Subject with contraindication for drawing blood
* Subject with medical pathology contraindicating sport practice
* Subject under treatments or drugs in the list of products prohibited for sports practice and competitions, in particular erythropoeitins and erythropoiesis-stimulating agents (updated list of World Anti-Doping Agency https://www.wada-ama.org/fr/liste-des-restrictions).
* Subject with physical or mental disability or restriction of liberty that would prevent autotransfusion
* Subject without a social security regimen
* Subject under guardianship or curatorship
* Subject participating in any Interventional study
* Positive HIV and/or hepatitis serology
* Discovery of a hematological disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  erythrocytes (/µL)
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  hemoglobin (g/dL)
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  Hematocrit (%)
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  Mean corpuscular volume (fL)
Change in hematological parameters | Baseline (Day 1), until 2 days after autotransfusion
  Reticulocyte by Sysmex analyzer
Variation in Red blood cells morphology | Baseline (Day 1), until 2 days after autotransfusion
  By amnis imaging flow cytometryProteins in Red blood cells (Wblot/ELISA/FACS)
Change in expression of cell surface proteins in red blood cells transfusion | Baseline (Day 1), until 2 days after autotransfusion
  Western blot /ELISA/ fluorescence-activated cell sorting of red blood cells
Change in microparticles detected in plasma | Baseline (Day 1), until 2 days after autotransfusion
  fluorescence-activated cell sorting

SECONDARY OUTCOMES:
Change in phthalate in urine | Baseline (Day 1), until 2 days after autotransfusion
  Assay by LC-MS/MS in urine

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HERMINE, MD, PhD, Principal Investigator — Assistance Publique-Hôpitaux Paris
Locations (1):
- EFS de Versailles, centre de soins, Le Chesnay-Rocquencourt, France

IPD SHARING:
Plan to Share IPD: No